CLINICAL TRIAL: NCT02458326
Title: Aerobic Training Effect on the Improvement of Pain Perception in Patients With Fibromyalgia and Migraine: a Randomized Clinical Trial
Brief Title: Aerobic Training Effect on the Improvement of Pain Perception in Patients With Fibromyalgia and Migraine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Manuella Moraes Monteiro Barbosa Barros, Physiotherapist, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37052114.3.0000.5208
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Migraine; Fibromyalgia
Keywords: Migraine; Fibromyalgia; Aerobic exercise
MeSH Terms: conditions — Migraine Disorders; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training (Experimental): The experimental group will follow the protocol: performing heating for 5 minutes at low speed on a treadmill; after heating, the speed is increased gradually until the patient reaches the proper heart rate for aerobic training obtained during cardiopulmonary exercise testing, maintaining the same for 20 minutes to perform the aerobic workout; completed, the velocity will be decreased to regain speed heating maintained for 5 minutes and finishing training. It is envisaged that in practice using the FC to ensure proper aerobic exercise for 20-60 minutes at a frequency of 3-5 times per week are effective in increasing the functional capacity of individuals with low fitness
  Interventions: Other: Aerobic training
- Control Training (Other): In the control group, these women will be guided to perform 10 minutes of heating on the treadmill with a low speed that does not cause patient effort (monitored by the Borg scale and FC close to the basement).
  Interventions: Other: Control Training

INTERVENTIONS:
Other: Aerobic training — Treadmill training with proper heart rate for aerobic workout to 20 minutes duration and frequency of three times a week for three months.
  Arms: Aerobic Training
Other: Control Training — 10 minutes of heating on the treadmill with a low speed that does not cause patient effort
  Arms: Control Training

SUMMARY:
Fibromyalgia and migraine are diseases with high prevalence in women between the age group of 30-60 years, which seem to share the same pathophysiological mechanism; both originate from neuroendocrine disorders of the hypothalamic-pituitary axis in the central nervous system, and are therefore closely related. In addition to the strong relationship with migraine, fibromyalgia can also be associated with sleep disorders, chronic fatigue and psychological disorders. The combination of these factors decreases the quality of life and contributes to increased sedentary this population. It is known that physical exercise promotes positive changes in pain pathophysiological pathway to increase the release of endorphins neuroendógenas, improving the symptoms of fibromyalgia.

The objective of this study is to analyze whether the application of an aerobic exercise program may result in the reduction of the frequency, duration and intensity of migraine attacks in women with fibromyalgia. For this, a clinical trial will be conducted randomized double-blind clinical trial comparing two groups of women diagnosed with fibromyalgia and migraine. Initially, all answer questionnaires assessing quality of life, impact of headache, level of depression and anxiety, sleep quality, physical activity level, and; will be held ergospirometry for research in exercise tolerance. The experimental group will implement the protocol consists of heating, aerobic exercise according to the heart rate established for training by spirometry and slowdown; and the control group will hold the heat on low speed and heart rate will next baseline. Both groups will be followed for 12 weeks, with a frequency of three weekly meetings lasting 30 minutes and re-evaluated every 4 weeks. At the end of the protocol, the groups will have their results were compared and statistically analyzed.

DETAILED DESCRIPTION:
This study is classified as a randomized double-blind clinical trial. Will be held in the Department of Physiotherapy of the university clinic of the Federal University of Pernambuco, located in University City, Recife-PE. Data for the survey will be collected during the course of the Masters in Physiotherapy, from April 2015 to September 2015, for further analysis.

The analyzed groups shall consist of women aged 30-50 years referred to the Department of Physical Therapy - UFPE, with clinical diagnosis of fibromyalgia and migraine performed by doctors of Rheumatology clinics and Neurology, Hospital das Clinicas, UFPE. Being invited to participate and informed about its content, saying their participation by signing a Term of Consent. Data collection is in accordance with the Declaration of Helsinki, and will begin after the project was approved by the Ethics Committee for Research on Human beings of the Federal University Health Sciences Center of Pernambuco, in accordance with Resolution 466/2012 of the National Research Ethics Committee of the Ministry of Health, the body that regulates research involving human subjects. The study will be registered in the digital Clinical Trials platform after obtaining the registration number of the Ethics Committee. Initially there will be a pilot study with 20 women, then the results will be used to calculate the sample size using the G Power (version 3.1.9.2, Germany), considering a statistical power (β) of 80% with a significance level (α) of 5%.

Will be excluded those that have some other rheumatologic disease, cardio-respiratory or cardiovascular that prevents the realization of aerobic exercise protocol; low attendance during the implementation of the exercise program (over three consecutive absences); cognitive impairment or neurological disease that compromises the understanding and the exercises; Body mass index ≥ 30.0 (obesity, according to the World Society of Health); pregnant women and patients classified as level of active or very active physical activity by IPAQ (International Physical Activity Questionnaire).

3.1. Randomization

Initially, patients will undergo will a simple randomization through the site www.randomization.com, resulting in two groups:

1. Aerobic Training: Submitted to a protocol consisting of heating, aerobic training with adequate heart rate and slowdown;
2. Control Training: Heating Protocol with speed and low intensity (heart rate will next basal).

Randomization will be performed by an examiner A, not research participant to ensure allocation concealment (patients and principal investigator will not be aware of which group are allocated). All women will be evaluated (both groups) through questionnaires and spirometry before the start and the end of the exercise protocol. Every four weeks, the patients will be submitted to revaluations through the questionnaires. The evaluation of these volunteers will be conducted by an examiner B (principal investigator), blinded to randomization; and the exercise protocol implementation will be the responsibility of the examiner C, only one will know to which group the patients belong. Corroborating the double-blinding, the evaluator to perform statistical analysis of the data will not know to which group belongs the results.

3.2. Evaluation

* Socio-demographic questionnaire Prepared by the researcher to characterize the groups, which answer questions for identification and history (name, date of valuation, telephone, address, date of birth, age, weight, height, body mass index / BMI, profession, education, marital status, physical activity and frequency, use of medication, type of medication, medication time). One minunciosa history regarding the use of drugs will be held: types, frequency, duration of treatment.
* Identification of the impact of migraine Will be evaluated by the Migraine Disability Assessment Test (MIDAS), which contains five items that measure the amount of days lost in the activities of daily living (ADLs) and professional (AVPs) due to the presence of migraine in the last three months; the patient declares the amount of days and, from the result of the sum of the scores, ranks the degree of disability of the individual (0-5 points: grade I / minimal disability; 6-10 points: grade II / mild disability; 11-20 points: grade III / moderate disability;> 20 points: grade IV / severe disability).
* Clinical characteristics of the headache Will be filled the journal Headache, based on criteria established by the International Headache Society (ICHD-III beta version, 2013); assesses the amount and duration of migraine attacks over a period of 30 days, pain intensity, symptoms associated with headache, medication use.
* Investigation of sleep quality The Pittsburgh Sleep Quality Index (PSQI), used to measure the subjective quality of sleep; consists of 19 items divided into seven components that punctuate 0-3 (total score of 0-21 points, the higher the score, the worse the quality of sleep). Was adapted and validated for the Brazilian population by Bertolazi and colleagues (2011), with a high reliability (α Cronbach = 0.82).
* Quality of life assessment Measured by the FIQ (Fibromyalgia Impact Questionnaire), consisting of 19 questions divided into 10 items: the first item has 10 sub-items with four response options ranging from 0-4 points; the second and third items, the patient should choose an option on a scale of 0-7; in the other, is given a score of 0-10 in response (the higher the score, the greater the impact of fibromyalgia on quality of life). Adapted and validated for the Brazilian population.
* Tracking of symptoms of anxiety and depression The presence of depression will be assessed by the Beck Depression Inventory (BDI), consisting of 21 questions that add up to a maximum score of 63 points (level of depression: 0-9 points = No; 10-18 points = mild depression; 19- 29 points = moderate depression;> 30 points = severe depression). It is validated and adapted for the Brazilian population, with a Cronbach's alpha of 0.81. The Beck Anxiety (BAI) will be used to identify and classify anxiety; consists of 23 statements that have the maximum score of 63 (0-10 points: minimum Anxiety, 11-19 points: Light Anxiety, points 20-30: moderate anxiety,> 31 points: severe anxiety), is validated and adapted to Brazilian population.
* Evaluation of the level of physical activity Proposed by the World Health Organization (1998), the International Physical Activity Questionnaire (IPAQ) aims to measure the total physical activity level (AFT) from the energy expenditure (METs.min-¹). Will be used to short IPAQ (version 8), which consists of 4 questions with two sub-items (b) on activities of daily living, professional life activities and practice of walking; where the frequency and duration respond if (days and hours / minutes) of activities and its intensity (moderate or vigorous = 3.3-4 METs = 5.5 to 8 METs) for one week. From the data obtained, sum up the frequency and duration of activities (walk + moderate + vigorous intensity) and, from this result, classifies individuals in: sedentary; irregularly active; active or very active. This questionnaire is validated and adapted for the Brazilian population, with excellent reproducibility (ICC = 0.79).
* Assessment of exercise tolerance Ergospirometry or cardio-pulmonary function test assesses precisely, the cardio-respiratory capacity and metabolic by direct measurement of maximum oxygen consumption and determining the maximum ventilatory thresholds. He is currently considered the gold standard for evaluation of exercise tolerance by providing non-invasive and very precise exercise intensities featuring aerobic or anaerobic metabolism (anaerobic threshold - LA). It is the most appropriate test for prescription of aerobic exercise intensity in sedentary individuals or with regular physical activity. Oxygen consumption (VO2 max) appears to be the most accurate indicator of exercise capacity. The test will be performed on a treadmill, coupled with a spirometer and a computer system in a climatically standardized environment. To minimize air leakage, will be employed the use of face masks with tiny dead-space. The main parameters obtained in the test are the ventilatory thresholds: anaerobic threshold (AT) and respiratory compensation point, which will characterize the aerobic and anaerobic workouts. The variables obtained during the test, with clinical relevance are: maximal oxygen uptake (VO2 max), carbon dioxide release (VCO 2), rate of gas exchange (R), estimated lactate threshold, expired minute volume (VE) , ventilatory reserve (RVE), ventilatory equivalents, end-expiratory pressures (PEF), ventilatory pattern, arterial gas tensions / oxyhemoglobin saturation, physiological dead space, electrocardiograms, heart rate, peripheral O2 saturation (SpO2) and blood pressure (BP ).

The responses to the cardiopulmonary exercise testing (CPX) are obtained by means of an incremental protocol, which consists in progressive load increases at predetermined time periods. A typical incremental protocol should provide: a resting phase (2-3 minutes or more), in which we observe a lack of hyperventilation before starting the test; a heating period with zero charge (2-3 minutes); incrementing a time (8-12 minutes) and an active period of recovery with no load (3-6 minutes if possible). For the intervention protocol, heart rate obtained just below the anaerobic threshold, recommended for proper intensity to gain fitness with greater security and compliance will be used. Generally, oxygen consumption levels in the anaerobic threshold are lower in these patients.

-Re-Reviews Initially, will be held the evaluation of patients through questionnaires and cardiopulmonary stress test to investigate exercise tolerance before the start of exercise protocol (review 1). Every 4 weeks, the patients of both groups will be reassessed by the re-application of all questionnaires: 4 weeks - review 2; 8 weeks: evaluation 3. At the end of the 12 weeks of training, the review 4 will be held, with repetition of the questionnaires and cardiopulmonary exercise testing.

3.3. Intervention protocol The intervention protocol will be made by the examiner C, one who is not blind to the research. After randomization and evaluation, patients will be allocated to one of the groups: experimental or control. After the evaluation of cardiorespiratory capacity of patients, will be established starting parameters appropriate to the level of physical activity each based on heart rate obtained just below the anaerobic threshold (ensuring aerobic work).

The experimental group will follow the following protocol: performing heating for 5 minutes at low speed on a treadmill; after heating, the speed is increased gradually until the patient reaches the proper heart rate for aerobic training obtained during cardiopulmonary exercise testing, maintaining the same for 20 minutes to perform the aerobic workout; completed, the velocity will be decreased to regain speed heating maintained for 5 minutes and finishing training. It is envisaged that in practice using the FC to ensure proper aerobic exercise for 20-60 minutes at a frequency of 3-5 times per week are effective in increasing the functional capacity of individuals with low fitness (American College of Sports Medicine - ACSM, 2006). In the control group, these women will be guided to perform 10 minutes of heating on the treadmill with a low speed that does not cause patient effort (monitored by the Borg scale and FC close to the basement).

Both groups will be followed for 12 weeks, with a driving frequency of 3 times per week. Heart rate and saturation of peripheral oxygen (SpO2) will be continuously monitored through the use of finger pulse oximeter during the course of all practices of all the volunteers of research to ensure that HR is within the established for each group

ELIGIBILITY:
Inclusion Criteria:

* Female
* 30-55 years
* Clinical diagnosis of fibromyalgia, according to the American College of Rheumatology criteria (2010)
* Migraine presence, according to the criteria of the International Headache Society (ICHD-III beta version, 2013).

Exclusion Criteria:

* Any other rheumatologic disease, cardio-respiratory or cardiovascular which prevents the realization of aerobic exercise protocol.
* Low attendance during the implementation of aerobic exercise protocol (over three consecutive fouls).
* Cognitive impairment or neurological disease that affects the understanding and the exercises.
* Pregnants
* Body mass index ≥ 30.0 (obesity, according to the World Health Company)
* Patients classified with level of active or very active physical activity by IPAQ (International Physical Activity Questionnaire)

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (headache) | End of aerobic exerise protocol (in the end of 12 weeks of training)
  At the end of the experimental protocol, it is expected that the intensity of migraine pain is reduced. Reviewed by MIDAS and headache diary.

SECONDARY OUTCOMES:
Duration of attacks of migraine | End of aerobic exerise protocol (in the end of 12 weeks of training)
  At the end of the experimental protocol, it is expected that the duration of attacks of migraine is reduced (days, hours). Reviewed by MIDAS and headache diary.
Frequence of migraine attacks | End of aerobic exerise protocol (in the end of 12 weeks of training)
  t the end of the experimental protocol, it is expected that the frequence of attacks of migraine is reduced (per months). Reviewed by MIDAS and headache diary.

CONTACTS AND LOCATIONS:
Overall Officials: Manuella MB Barros, Master, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil